CLINICAL TRIAL: NCT05859776
Title: Phase 1/2a Study of the Safety and Bioactivity of AXT107 Injected Suprachoroidally in Subjects With Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: Safety and Bioactivity of AXT107 in Subjects With Neovascular Age-Related Macular Degeneration (nAMD)
Acronym: DISCOVER
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AsclepiX Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AXT107-CS104
Record Dates: First submitted 2023-03-24; First posted 2023-05-16 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — AXT107

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): AXT107 0.125 mg/eye
  Interventions: Drug: AXT107 Low Dose
- Mid Dose (Experimental): AXT107 0.250 mg/eye
  Interventions: Drug: AXT107 Mid Dose
- High Dose (Experimental): AXT107 0.500 mg/eye
  Interventions: Drug: AXT107 High Dose

INTERVENTIONS:
Drug: AXT107 Low Dose — Single suprachoroidal injection of AXT107 (0.125 mg/eye)
  Other Names: Gersizangatide
  Arms: Low Dose
Drug: AXT107 Mid Dose — Single suprachoroidal injection of AXT107 (0.250 mg/eye)
  Other Names: Gersizangatide
  Arms: Mid Dose
Drug: AXT107 High Dose — Single suprachoroidal injection of AXT107 (0.500 mg/eye)
  Other Names: Gersizangatide
  Arms: High Dose

SUMMARY:
The goal of this clinical trial is to understand the safety of AXT107 injected suprachoroidally in participants with nAMD. The main question[s] it aims to answer are:

* Safety of the maximum tolerable dose of AXT107
* Bioactivity and duration of action of AXT107 injected suprachoroidally Participants will be injected with AXT107 and will be followed on a regular monitoring visits through 9 months post single injection.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Presence of active subfoveal choroidal neovascularization (CNV) (any subtype) or juxtafoveal CNV with leakage affecting the fovea secondary to AMD and the area of the CNV lesion must beat least 50% of the total lesion size confirmed by the Investigator
* Evidence of subretinal or intraretinal fluid or retinal cystic changes evidenced by Spectral Domain Optical Coherence Tomography (SD-OCT) at Screening accompanied by finding on SD- OCT suggestive of CNV secondary to AMD confirmed by the Investigator
* BCVA in the study eye between 65 and 25 ETDRS letters (20/50 and 20/320 Snellen equivalent) at Baseline (Day 0)
* BCVA of 34 ETDRS letters or better (20/200 or better Snellen equivalent) in the non-study eye at Baseline (Day 0)
* Able and willing to give signed informed consent and follow study instructions
* Has been/is a prior partial responder to an anti-VEGF agent

Exclusion Criteria:

* Previously treated patients who are non-responders to anti-VEGF as determined by the Investigator
* Any prior use of Brolucizumab; use of Aflibercept within 8 weeks or use of Ranibizumab or Bevacizumab within 6 weeks from Baseline (Day 0) in the study eye
* Any concurrent disease that would require medical or surgical intervention during the study in the study eye (e.g., retinal detachment, significant cataract)
* Any condition that may preclude improvement in visual acuity or affect the evaluation of the study eye after resolution of AMD (e.g., extensive macular hemorrhage ≥ 50% lesion size, media clarity insufficient to obtain quality images, presence of diabetic retinopathy)
* Other causes of CNV (e.g., pathologic myopia, ocular histoplasmosis syndrome, angioid streaks, and multifocal choroiditis) in the study eye confirmed by the Investigator
* Chronic uveitis or ongoing clinically significant infection or inflammation (e.g., keratitis, scleritis) in either eye

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 40 Weeks
  Primary Outcome Measure:
  1.Safety as Assessed by change from baseline in Incidence of Adverse Events (AEs) Incidence of ocular (study eye) and systemic AEs
  [Time Frame: Screening to Week 40]

SECONDARY OUTCOMES:
Mean Change in Central Subfield Thickness (CST) | 40 Weeks
  Secondary Outcome Measures:
  Efficacy as Assessed by Central Subfield Thickness (CST, measured in µm) Mean change in CST assessed by spectral domain optical coherence tomography
  [Time Frame: Day 0 to Week 40]
Mean Change in Visual Function | Day 0 to Week 40
  Secondary Outcome Measures:
  Visual Function as Assessed by Mean change in Best Corrected Visual Acuity (BCVA) (number of letters in Early Treatment Diabetic Retinopathy Study (EDTRS) chart)
Visual Function Subgroup Analysis | Day 0 to Week 40
  Secondary Outcome Measures:
  Visual Function as Assessed by Early Treatment Diabetic Retinopathy Study (EDTRS) Chart Percentage of subjects improving ≥5, ≥10, and ≥15 letters in Best Corrected Visual Acuity (BCVA)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - New England Retina Consultants, Springfield, Massachusetts
  - The Retina Institue, St Louis, Missouri
  - Asheville Eye Associates, Asheville, North Carolina
  - Erie Retina Research, Erie, Pennsylvania

IPD SHARING:
Plan to Share IPD: No